CLINICAL TRIAL: NCT06136494
Title: Patient and Societal Benefits of Guided Internet-delivered Cognitive Behavioural Therapy for Cardiac Anxiety in Patients With Non-cardiac Chest Pain
Brief Title: iCBT for Cardiac Anxiety in Patients With NCCP
Acronym: IKSIT2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ghassan Mourad, Senior Associate Professor (Docent), Linkoeping University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: iCBT for NCCP
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Non-cardiac Chest Pain; Cardiac Anxiety
Keywords: Cardiac anxiety; Cognitive behavioural therapy; Internet-delivered; Noncardiac chest pain; Psychological distress; Cost-effectiveness; Therapeutic alliance

STUDY DESIGN:
Intervention Model Description: iCBT versus attention control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive an 8-week guided iCBT-program including goal setting, psychoeducation, physical activity, exposure, mindfulness, and acceptance.
  Interventions: Behavioral: Internet-delivered cognitive behavioural therapy
- Control group (Active Comparator): The control group will receive general support via weekly email contact to check how they are feeling and how they are dealing with their situation. The control group will be offered iCBT after 3 months.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioural therapy — Psychoeducation aims at teaching patients about chest pain and anxiety and their impact on daily life. Mindfulness is used to raise awareness of what is going on in the body and emotions and to learn how to relate to chest pain. Physical activity consists of psychoeducation and recommendations regarding physical activity with the goal to get patients to learn that their heart tolerates physical activity and to reduce cardiac anxiety and avoidance of physical activity. Avoidance/exposure is to teach patients how avoidance and safety behaviours can maintain/exacerbate chest pain and negatively impact daily life. Acceptance is about learning to accept having the chest pain without letting it take over one's life. The participants will have weekly assignments with weekly feedback and advice. Reminders and encouraging messages will be sent to motivate participants to complete the intervention. The treatment will be carried out through our own web platform.
  Other Names: iCBT
  Arms: Intervention group
Behavioral: Attention control — General support via weekly email contact to check how participants are feeling and how they are dealing with their situation. iCBT will be offered after 3 months.
  Arms: Control group

SUMMARY:
Non-cardiac chest pain (NCCP) is a common condition that significantly affects patients' mental well-being, overall quality of life, and healthcare use. Even after ruling out cardiac issues, many patients still worry about having an undiagnosed cardiac illness, leading to cardiac anxiety since no other explanation is provided. Consequently, they avoid activities they believe might harm their heart, worsening their overall health and resulting in increased healthcare visits and societal costs. Addressing cardiac anxiety through psychological interventions could help break this viscious cycle and enhance patient outcomes. Internet-delivered cognitive behavioural therapy (iCBT) can assist patients in reassessing their perceptions, emotions and behaviours in order to handle their chest pain and therby reduce their cardiac anxiety.

The aim of this study is to evaluate the short- and long-term effects of a guided 8-week iCBT program on cardiac anxiety, generalized anxiety, kinesiophobia, fear of body sensations, depressive symptoms, health-related quality of life, chest pain frequency and illness perception. Also to examine how participants' personality traits influence the effectiveness of the iCBT program. Furthermore, to assess the cost-effectiveness of the iCBT program compared to attention control. In addition, we will explore the perceptions of participants regarding the therapeutic alliance during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* experience of non-cardiac chest pain
* exhibiting cardiac anxiety (score ≥24 on the Cardiac Anxiety Questionnaire, CAQ)

Exclusion Criteria:

* language difficulties
* patients with no access to computer/tablet and/or Internet
* not able to perform physical activity/exercise due to physical constraints
* severe psychological disorders or chronic somatic illness assessed to be requiring acute treatment or to hinder participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac Anxiety | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  Cardiac Anxiety Questionnaire (CAQ) will be used to assess the short- and long-term effects of the intervention on cardiac anxiety. The CAQ consists of 18 items and a score range between 0 and 72. The higher scores the greater cardiac anxiety.

SECONDARY OUTCOMES:
Generalized anxiety | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  The Generalized Anxiety Disorder 7 (GAD-7) will be used to assess the severity of symptoms in individuals experiencing anxiety. It consists of 7 items with scores ranging between 0 and 21 with higher scores indicating more severe anxiety symptoms.
Kinesiophobia | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  The Tampa Scale for Kinesiophobia (TSK) will be used to assess the fear of movement. It consists of 17 items that measure various aspects of kinesiophobia, including avoidance behaviour and the belief that movement may cause harm. Scores range between 17 and 68, with higher scores indicating a higher level of fear of movement.
Fear of body sensations | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  Body Sensations Questionnaire will be used to assess fear of body sensations. The questionnaire comprises 17 items with scores ranging between 17 and 85 and the higher scores the greater fear of body sensations.
Depressive symptoms | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  Patient Health Questionnaire-9 will be used to assess changes in depressive symptoms related to intervention. This questionnaire comprises 9 items with scores ranging between 0 and 27. Higher scores indicate higher levels of depressive symptoms.
Health-related quality of life | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  EuroQol-5D (EQ-5D) includes five dimensions of Health-related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels corresponding to: no problems, slight problems, moderate problems, severe problems and extreme problems/unable. The questionnaire also includes an EQ-VAS, which is a visual analogue scale ranging from 0 (worst health you can imagine) to 100 (best health you can imagine).
Chest pain prevalence | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  Self-developed open questions will be used to asses the frequency and intensity of perceived chest pain.
Illness perception | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  The Revised Illness Perception Questionnaire (IPQ-R) is designed to assess individuals' perceptions and beliefs about their illness or health condition, i.e. NCCP. It evaluates various components, such as their understanding of the illness, perceived consequences, timeline, personal control, treatment control, and emotional representations related to the illness. The questionnaire helps to understand patients' cognitive and emotional representations of their health condition, which can influence their coping strategies and health-related behaviours.
Personality traits | Measurements will be performed before and after the intervention (8 weeks), and 3, 6, 12, and 24 months after the end of the intervention.
  The Ten-Item Personality Inventory (TIPI) is used to assess an individual's personality traits. It consists of ten items, with two items for each of the Big Five personality traits: extraversion, agreeableness, conscientiousness, emotional stability (or neuroticism), and openness to experience. Participants rate themselves on a scale from 1 to 7 for each item, indicating the extent to which they agree or disagree with the statements.
Healthcare use | Data will be collected one year prior to and one year post intervention
  In-patient (hospital admissions and length of stay, and outclinic visits at hospital), and out-patient data (primary care visits/consultations) will be collected frpom data care registries.
Healthcare costs | Data will be collected one year prior to and one year post intervention
  Healthcare costs will be collected from cost registers.

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Mourad, Principal Investigator — Department of Health, Medicine and Caring Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No